CLINICAL TRIAL: NCT04717206
Title: Effects of 6 Weeks Plyometric Training on Vertical Jump and Agility in Relation to Gender Among Badminton Players
Brief Title: 6 Weeks Plyometric Training on Vertical Jump and Agility in Relation to Gender Among Badminton Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/717 Shakeela Parveen
Record Dates: First submitted 2020-11-11; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Sports Physical Therapy
Keywords: Strength Training; Plyometric training; Agility; Vertical Jump

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyomtric training to male badmninton players (Experimental): Baseline assessment will be perfomimg on first day before intervention, 4 weeks plyometric training to male badminton players.
  Interventions: Other: Plyomtric training to male badmninton players
- Plyomtric training to female badmninton players (Experimental): Baseline assessment will be perfomimg on first day before intervention, 4 weeks plyometric training to female badminton players.
  Interventions: Other: Plyomtric training to female badmninton players

INTERVENTIONS:
Other: Plyomtric training to male badmninton players — Plyometric training has been proven to be effective and effecient in developing strength and speed.
  plyometric training includes different types hops,jumping,drills.
  Arms: Plyomtric training to male badmninton players
Other: Plyomtric training to female badmninton players — Plyometric training has been proven to be effective and effecient in developing strength and speed.
  plyometric training includes different types hops,jumping,drills.
  Arms: Plyomtric training to female badmninton players

SUMMARY:
This study exmine the effects of plyometric training on vertical jump and agility in male and female badminton players.The two groups will be subsequently randomly assign into the experimental group and control group.

DETAILED DESCRIPTION:
After approval from the graduate committee permission will be obtained from the higher authorities of the naval anchorage badminton club islamabad. Purpose of this study will be explained to the all participants written informed consent will be obtained.participants will recive 6 weeks intervention with a generic warm up consisting of ten body weight squats,ten forward lunges each side and 3 mintues of dynamic stretching of relevant lower extremity muscles. The agility t-test will be used to measure and seargent vertical jump test will be used to measure vertical jump.

ELIGIBILITY:
Inclusion Criteria:

* Male and female clients
* Players whose age lies between 18 and 25 years.
* Players who played badminton for at least 6 months

Exclusion Criteria:

* Musculoskeletal or neurological disease
* Pathological condition of spine , hip, knee and pelvic

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Agility T-test | 6 to 8 weeks
  The T-Test is a simple running test of agility, involving forward, lateral, and backward movements, appropriate to a wide range of sports.
  Equipment required: marker cones, measurement tape, stopwatch, non-slip surface.
  Pre-test: Explain the test procedures to the subject. Perform screening of health risks and obtain informed consent. Prepare forms and record basic information such as age, height, gender, test conditions. Measure and mark out the test area. Perform an appropriate warm-up.
  Procedure: The subject starts at cone A. On the command of the timer, the subject sprints to cone B and touches the base of the cone with their right hand. They then turn left and shuffle sideways to cone C, and also touches its base, this time with their left hand. Then shuffling sideways to the right to cone D and touching the base with the right hand. They then shuffle back to cone B touching with the left hand, and run backwards to cone A. The stopwatch stopped as they pass cone A
Vertical Jump Test (Sargent Jump) | 6 to 8 weeks
  This test is designed to measure lower limb explosive power by measuring the height a client is able to jump.
  Equipment required: measuring tape, chalk for marking wall Description / procedure: The person stands side on to a wall and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked or recorded. This is called the standing reach. The person puts chalk on their fingertips to mark the wall at the height of their jump. The person then stands away from the wall, and jumps vertically as high as possible using both arms and legs to assist in projecting the body upwards. Attempt to touch the wall at the highest point of the jump. The difference in distance between the standing reach height and the jump height is the score. The best of three attempts is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Karim, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Naval Anchorage badminton club, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Villarreal ES, Kellis E, Kraemer WJ, Izquierdo M. Determining variables of plyometric training for improving vertical jump height performance: a meta-analysis. J Strength Cond Res. 2009 Mar;23(2):495-506. doi: 10.1519/JSC.0b013e318196b7c6. PMID 19197203
- [Background] Alikhani R, Shahrjerdi S, Golpaigany M, Kazemi M. The effect of a six-week plyometric training on dynamic balance and knee proprioception in female badminton players. J Can Chiropr Assoc. 2019 Dec;63(3):144-153. PMID 31988535
- [Background] Khodami A, Nikseresht A, Khoshnam E. The effect of 8 weeks of plyometric training on cortisol and DHEA Levels in male badminton players. Eur J Exp Biol. 2014;4(1):265-9.
- [Background] Sozbir K. Effects of 6-week plyometric training on vertical jump performance and muscle activation of lower extremity muscles. US Sports Academy. 2016.
- [Background] Irawan D, editor Six Weeks Progressive Plyometrics Training on Badminton Player's Agility. Health Science International Conference (HSIC 2017); 2017: Atlantis Press.
- [Background] Kashmira S, Seema S. Comparison between depth jump and counter-movement jump for increasing vertical jump height in male Badminton players. Journal of Orthopaedics and Rehabilitation. 2011;1(1).
- [Background] Voisin MPJ, Scohier M. Effect of an 8-Week Plyometric Training Program with Raised Forefoot Platforms on Agility and Vertical Jump Performance. Int J Exerc Sci. 2019 Mar 1;12(6):491-504. doi: 10.70252/FNWU6350. eCollection 2019. PMID 30899356
- [Background] OZMEN T, AYDOGMUS M. Effect of plyometric training on jumping performance and agility in adolescent badminton players. Turkish Journal of Sport and Exercise. 2017;19(2):222-7.
- [Background] Harvey C. The relationship between jump testing in badminton and on-court jumping drills in elite badminton players: University of Wales Institute Cardiff; 2010.
- [Background] McNellie T. THE EFFECTS OF A SIX WEEK PLYOMETRIC TRAINING PROGRAMME ON THE AGILITY OF MALE CRICKETERS. 2013.
- [Background] Raya MA, Gailey RS, Gaunaurd IA, Jayne DM, Campbell SM, Gagne E, Manrique PG, Muller DG, Tucker C. Comparison of three agility tests with male servicemembers: Edgren Side Step Test, T-Test, and Illinois Agility Test. J Rehabil Res Dev. 2013;50(7):951-60. doi: 10.1682/JRRD.2012.05.0096. PMID 24301432
- [Background] Klavora P. Vertical-jump tests: A critical review. Strength and Conditioning Journal. 2000;22(5):70-5.